CLINICAL TRIAL: NCT07235384
Title: A Phase 1/1b Randomized, Double Blind, Placebo-controlled, Single and Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ZL-1503 in Healthy Volunteers and Participants With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: A Phase 1/1b Study to Evaluate Safety, Tolerability and Pharmacokinetics of ZL-1503 in Healthy Volunteers and Participants With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZL-1503-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZL-1503: Participants will receive single ascending doses of ZL-1503 (Experimental): Part A: Single Ascending Dose (SAD)
  Interventions: Drug: ZL-1503; Drug: Placebo
- ZL-1503: Participants will receive multiple ascending doses of ZL-1503 (Experimental): Part B: Multiple Ascending Dose (MAD)
  Interventions: Drug: ZL-1503; Drug: Placebo

INTERVENTIONS:
Drug: ZL-1503 — Healthy volunteers will receive ZL-1503.
  Arms: ZL-1503: Participants will receive single ascending doses of ZL-1503
Drug: Placebo — Healthy volunteers will receive placebo.
  Arms: ZL-1503: Participants will receive single ascending doses of ZL-1503
Drug: ZL-1503 — Participants with moderate to severe atopic dermatitis will receive ZL-1503.
  Arms: ZL-1503: Participants will receive multiple ascending doses of ZL-1503
Drug: Placebo — Participants with moderate to severe atopic dermatitis will receive placebo.
  Arms: ZL-1503: Participants will receive multiple ascending doses of ZL-1503

SUMMARY:
This is a phase 1/1b randomized, double blind, placebo-controlled, single dose escalation (SAD) and multiple dose escalation (MAD) study to evaluate the safety, tolerability, and pharmacokinetics (PK) of ZL-1503 in healthy volunteers and participants with moderate to severe atopic dermatitis (AD)

DETAILED DESCRIPTION:
The study consists of two parts:

* Part A: single ascending dose in healthy volunteers
* Part B: multiple ascending doses in adult participants with moderate to severe AD

ELIGIBILITY:
Inclusion Criteria:

* Part A:

  1. Healthy male and female volunteers, 18-65 years of age
  2. Body mass index (BMI) between ≥ 18.5 and < 32.5 kg/m2
  3. Negative pregnancy tests for women of childbearing potential.
* Part B:

  1. 18-65 years of age;
  2. BMI between ≥18.5 and <40.0 kg/m2
  3. Have a diagnosis of AD at least 12 months prior to Day 1;
  4. Moderate-to-severe AD at Screening and Baseline visit, defined as:

     1. Eczema Area and Severity Index (EASI) score ≥ 16;
     2. Affected Body Surface Area (BSA)≥ 10%;
     3. vIGA-AD™ score ≥ 3
  5. History of an inadequate response to treatment with topical medications
  6. Average peak pruritus numeric rating scale (PP-NRS) score ≥4 in the 7 days before randomization.
  7. Negative pregnancy tests for women of childbearing potential.

Exclusion Criteria:

* Part A and B:

  1. Significant health issues, such as positive tests for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg), active tuberculosis, immunodeficiencies or autoimmune diseases.
  2. History of major metabolic, liver, kidney, hematologic or other significant disorders.
  3. Abnormal Electrocardiogram (ECG) findings
  4. Clinically relevant abnormal lab results, including low blood counts, or abnormal liver and kidney function.
  5. History of drug abuse or addiction within 6 months prior to screening
  6. Current smoker or use of any nicotine or tobacco containing products within the last 6 months prior to dosing.
  7. Donated >500mL blood within 2 months of dosing.
* For Part B only:

  1. Presence of dermatologic conditions and/or comorbidities that might confound the diagnosis of AD and/or might interfere with study assessments.
  2. Uncontrolled chronic disease that might require bursts of oral corticosteroids.
  3. Any other sound medical, psychiatric, and/or social reason as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 48 weeks after last intervention
Number of participants with serious adverse events (SAEs) | Up to 48 weeks after last intervention
Number of participants with clinical laboratory abnormalities | Up to 48 weeks after last intervention
Number of participants with vital sign abnormalities | Up to 48 weeks after last intervention
Number of participants with electrocardiogram (ECG) abnormalities | Up to 48 weeks after last intervention

CONTACTS AND LOCATIONS:
Locations (1):
- ZaiLab Site 18001, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No